CLINICAL TRIAL: NCT00774930
Title: A Double Blind, Randomized Placebo Controlled Clinical Trial Investigating the Efficacy and Safety of Somatuline Depot (Lanreotide) Injection in the Treatment of Carcinoid Syndrome
Brief Title: An Efficacy and Safety Study of Somatuline Depot (Lanreotide) Injection to Treat Carcinoid Syndrome
Acronym: ELECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-55-52030-730; TR321 (Other: Tercica Inc); 2010-019066-92 (EudraCT Number)
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-09

CONDITIONS: Carcinoid Syndrome
Keywords: Carcinoid tumor; Somatuline Depot; Lanreotide Autogel; Neuroendocrine tumor; NET; Diarrhea; Flushing; Carcinoid tumour; Neuroendocrine tumour; Diarrhoea
MeSH Terms: conditions — Serotonin Syndrome; Carcinoid Tumor; Neuroendocrine Tumors; Diarrhea; Flushing | interventions — lanreotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lanreotide Autogel (Somatuline Depot) 120 mg (Experimental): Subjects received deep s.c. lanreotide Autogel 120 mg every 4 weeks (±3 days) for 16 weeks (DB phase).
  After completing the DB phase (or if they met criteria for early roll over [ERO]) the subjects entered the IOL phase during which they received lanreotide Autogel 120 mg deep s.c. every 4 weeks for 32 weeks. During the LTOLE phase, subjects continued treatment with lanreotide Autogel 120 mg deep s.c. every 4 weeks until at least 2 years after the last subject completed the IOL phase or when marketing approval for the treatment of symptoms of carcinoid syndrome was obtained [whichever occurred first]).
  Interventions: Drug: Lanreotide
- Placebo (DB) and lanreotide Autogel 120 mg in IOL and LTOLE (Placebo Comparator): Subjects received deep s.c. placebo every 4 weeks (±3 days) for 16 weeks (DB phase).
  After completing the DB phase (or if they met criteria for ERO) the subjects entered the IOL phase during which they received lanreotide Autogel 120 mg deep s.c. every 4 weeks for 32 weeks. During the LTOLE phase, subjects continued treatment with lanreotide Autogel 120 mg deep s.c. every 4 weeks until at least 2 years after the last subject completed the IOL phase or when marketing approval for the treatment of symptoms of carcinoid syndrome was obtained [whichever occurred first]).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lanreotide — deep s.c. injection, 120 mg, every 4 weeks (±3 days).
  Other Names: Somatuline; Somatuline Depot; Somatuline Autogel; Lanreotide Autogel
  Arms: Lanreotide Autogel (Somatuline Depot) 120 mg
Drug: Placebo — deep s.c. injection of placebo (0.9% saline solution) every 4 weeks (±3 days) for 16 weeks, then deep s.c. injection of lanreotide 120 mg, every 4 weeks (±3 days).
  Arms: Placebo (DB) and lanreotide Autogel 120 mg in IOL and LTOLE

SUMMARY:
The purpose of this study was to determine whether monthly deep subcutaneous (s.c.) injections of lanreotide Autogel (Somatuline Depot) were effective and safe in controlling diarrhoea and flushing by reducing the usage of s.c. short-acting octreotide as a rescue medication to control symptoms in subjects with carcinoid syndrome.

DETAILED DESCRIPTION:
This study consisted of a Screening period, conducted up to 4 months before randomisation, followed by three phases: a 16-week, double blind (DB), randomised, placebo-controlled phase; a 32-week initial open label (IOL) phase; and a long term open label extension (LTOLE) phase.

The DB phase evaluated lanreotide Autogel versus placebo in subjects with a history of carcinoid syndrome (flushing and/or diarrhoea). This was followed by a 32-week IOL phase in which all subjects received lanreotide Autogel 120 mg every 4 weeks. Subjects in countries where lanreotide Autogel had not been approved for the treatment of carcinoid syndrome, who were well-controlled at the end of the 32-week IOL phase and chose to continue to receive lanreotide Autogel, were given the option of participating in a LTOLE phase. The LTOLE phase of the study was planned to end at least 2 years after the last subject had completed his/her participation in the 32-week IOL phase or when marketing approval for the treatment of symptoms of carcinoid syndrome had been obtained in the respective countries (whichever occurred first) or at any time the study was terminated by the Sponsor. The actual overall duration of the study was 6.5 years. During the LTOLE phase all subjects continued to be treated with lanreotide Autogel 120 mg every 4 weeks.

The study planned to enrol approximately 100 adult subjects worldwide. Screening continued until 115 subjects were enrolled in the study.

ELIGIBILITY:
Subjects were eligible for participation in the study if they met the following criteria:

1. At least 18 years of age at the time of first dosing.
2. Subjects must have given signed informed consent before any study related activities were conducted.
3. Subjects in the United States of America (USA) must have given written authorisation for the release of protected health information in compliance with the Health Insurance Portability and Accountability Act (HIPAA) regulations; subjects in other countries must have provided appropriate authorisation as needed by regulatory authorities in each country.
4. Subjects must have been willing to receive s.c. octreotide injections as rescue medication, as needed to control their symptoms, if any.
5. If female, the subject must not have been pregnant (confirmed by negative pregnancy test) and must have had the following documented via verbally given history:

   * At least 1 year postmenopausal (natural cessation of menses), or
   * Surgically sterile (if by tubal ligation, surgery must have been performed more than 3 months prior to entry into the study), or
   * If the subject was of childbearing potential and sexually active, she must have been using an acceptable form of contraception (oral, injected, transdermal or implanted contraceptives, diaphragm or barrier method with spermicidal and/or intrauterine device); local methods such as condoms or sponges/vaginal tablets were not acceptable forms of contraception.
6. Subjects with a histopathologically confirmed diagnosis of carcinoid tumour or, a carcinoid tumour of unknown location with liver metastases (documented biopsy), and a history of carcinoid syndrome (flushing and/or diarrhoea) who were either naïve to treatment with a somatostatin analogue (SSTa) or responsive (according to the opinion of the principal investigator) to conventional doses of Sandostatin LAR® Depot (LAR; ≤30 mg every 4 weeks) or to daily doses of ≤600 μg of s.c. octreotide.
7. Confirmation of positive somatostatin receptor (SSTR) status by somatostatin receptor scintigraphy (SRS; up to 6 months prior to study entry at the Screening Visit).
8. Absence of tumour progression documented by two sequential computed tomography (CT) scans or two sequential magnetic resonance imaging (MRI) scans (≥3 months apart); the last CT or MRI scan must have been performed within 6 months of study entry (Screening Visit).
9. Subjects previously treated with LAR, must have received their last dose of LAR at least 4 weeks prior to first dose of study treatment (no later than at the Screening Visit).
10. Be able to communicate and cooperate with the principal investigator and the staff and willing to comply with the study instructions.

Subjects were excluded from entering the study for the following reasons:

1. History of known allergy or hypersensitivity to investigational drug or any components of its formulation, or octreotide.
2. History of carcinoid syndrome refractory to treatment with conventional doses of SSTa.
3. Treatment with any other investigational drug within 30 days prior to study entry (Screening Visit) and/or at any time during the subject's participation in the study.
4. Treatment with interferon, chemotherapy and/or radiotherapy (a radiolabelled SSTa) and/or tumour debulking <3 months prior to study entry (Screening Visit).
5. History of hepatic arterial embolisation, hepatic arterial chemoembolisation and/or selective internal radiation therapy (selective internal radiation [SIR] therapy [SIRT]; e.g. SIR Spheres) <6 months prior to study entry (Screening Visit).
6. Short bowel syndrome.
7. Uncontrolled diabetes and/or hypertension.
8. Severe renal impairment (glomerular filtration rate <30 mL/min/1.73 m2) and/or severe liver impairment as evidenced by serum total bilirubin >1.5 mg/dL associated with bile duct blockage or with alkaline phosphatase (ALP), aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5.0 upper limit of normal (ULN).
9. Diagnosis of cardiac disease New York Heart Association (NYHA) functional classification >Class I. (Subject has limitation of physical activity. Ordinary physical activity causes undue fatigue, palpitation, or dyspnoea).
10. Life expectancy less than 1 year.
11. Any malignancies except carcinoid tumour, basocellular carcinoma of the skin, in situ carcinoma of the cervix and ≥5 years disease free after curative cancer treatment.
12. Any serious medical condition that could jeopardise the safety of the subject and/or the efficacy assessments of the study.
13. Subject is being treated with a proton pump inhibitor (PPI) and has been at a stable dose (no change in dose or frequency of administration) for less than 4 weeks at study entry (Screening Visit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-05; Primary Completion 2013-05 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (54):
- United States (16):
  - VA Greater Los Angeles Health Care System, Los Angeles, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Stanford Cancer Center, Stanford, California
  - Cedars Sinai Outpatient Cancer Center, West Hollywood, California
  - Kentuckiana Cancer Institute, Louisville, Kentucky
  - Louisiana State University Health Science Center, Kenner, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of New Mexico Cancer Care Center, Albuquerque, New Mexico
  - Providence Portland Medical Center, Portland, Oregon
  - Oregon Health Science University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Liver Cancer Center, Pittsburgh, Pennsylvania
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin
- Brazil (7):
  - Biocancer - Centro de Pesquisa e Tratamento do Câncer, Belo Horizonte
  - Hospital LifeCenter, Belo Horizonte
  - Oxion Medicina Oncológica, Belo Horizonte
  - Hospital Universitário de Brasilia, Brasília
  - Hospital Erasto Gaertner, Curitiba
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Hospital de Base de São José do Rio Preto, São José do Rio Preto
- VFN Onkologicka klinika, Prague, Czechia
- India (7):
  - Sir Gangaram Hospital, Delhi
  - Indo-American Cancer Institute & Research Centre, Hyderabad
  - Omega Hospitals, Hyderabad
  - Santokaba Durlabhji Memorial Hospital and Research Institute, Jaipur
  - Bhagwan Mahaveer cancer hospital and research centre, Jaipur
  - Shatabdi Super Speciality hospital, Mumbai
  - Tata Memorial Hospital, Mumbai
- Paul Stradins Clinical University Hospital, Riga, Latvia
- Klinika Endokrynologii, Diabetologii i Leczenia Izotopami, Wroclaw, Poland
- Russia (3):
  - Non-Federal Institution of Healthcare "Central Clinical Hospital # 1 of the LLC "Russian Railways (RZD)", Moscow
  - Russian Academy of Medical Sciences "Russian Oncological Research Centre named after N.N. Blokhin RAMS", Moscow
  - Federal Institution of Healthcare "Leningradsky Regional Oncological Dispensary", Saint Petersburg
- Serbia (2):
  - Clinic of Endocrinology, diabetes and metabolic diseases, Clinical Center of Serbia, Belgrade
  - Oncology Institute of Vojvodina, Sremska Kamenica, Kamenitz
- South Africa (4):
  - Rondebosch Oncology Unit, Cape Town
  - Groote Schuur Hospital, Cape Town
  - Westridge Medical Centre, Durban
  - GVI Oncology Clinical Trial Unit, Port Elizabeth
- Erciyes University Medical Faculty, Kayseri, Turkey (Türkiye)
- Ukraine (11):
  - Cherkassy Regional Oncology Dispensary, Cherkassy
  - Chernivtsi Regional Oncology Center, Chernivtsi
  - Oncology and Medical Radiology Chair of Dnepropetrovsk State Medical Academy, Dnipro
  - Regional Anticancer Center, Department of oncoproctology, Donetsk
  - Municipal Clinical Hospital #2, Proctology department, Kharkiv
  - Kyiv City Oncological Hospital, Thoracic department, Kyiv
  - Medical Centre "Mriya", Kyiv
  - National Cancer Institute, Kyiv
  - Odessa Regional Clinical Hospital, Odesa
  - Uzhgorods'ka Tsentral'na Mis'ka Klinichna Likarnya, Mis'kyy Onkologichnyy Tsentr, Uzhhorod
  - Vinnytsya Regional Clinical Oncological Center, Vinnytsya State Medical University, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Result] Vinik AI, Wolin EM, Liyanage N, Gomez-Panzani E, Fisher GA; ELECT Study Group *. EVALUATION OF LANREOTIDE DEPOT/AUTOGEL EFFICACY AND SAFETY AS A CARCINOID SYNDROME TREATMENT (ELECT): A RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED TRIAL. Endocr Pract. 2016 Sep;22(9):1068-80. doi: 10.4158/EP151172.OR. Epub 2016 May 23. PMID 27214300
- [Derived] Blot K, Duchateau L, Lescrauwaet B, Liyanage N, Ray D, Mirakhur B, Vinik AI. A Patient-Reported Outcomes Analysis Of Lanreotide In The Treatment Of NETs Patients With Carcinoid Syndrome: Evidence From The ELECT Trial. Patient Relat Outcome Meas. 2019 Oct 29;10:335-343. doi: 10.2147/PROM.S219982. eCollection 2019. PMID 31754316

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from multiple sites across countries from May 2009. The study was completed in December 2015.
Pre-assignment Details: A total of 153 subjects were screened; 115 were randomized and 38 failed screening.
Groups:
- Lanreotide Autogel (Somatuline Depot) 120 mg: Deep s.c. injections of lanreotide Autogel 120 mg every 4 weeks (±3 days) for 16 weeks (DB phase). Subjects then received deep s.c. injections of lanreotide Autogel 120 mg every 4 weeks for 32 weeks in the initial open label (IOL) phase and further deep s.c. injections with lanreotide Autogel every 4 weeks in the long term open label extension (LTOLE) phase.
- Placebo: Deep s.c. injections of placebo every 4 weeks (±3 days) for 16 weeks (DB phase). Subjects then received deep s.c. injections of lanreotide Autogel 120 mg every 4 weeks for 32 weeks in the IOL phase and further deep s.c. injections with lanreotide Autogel every 4 weeks in the LTOLE phase.
Period: DB Phase
Arm/Group | Lanreotide Autogel (Somatuline Depot) 120 mg | Placebo
Started | 59 (One subject was randomised to receive lanreotide Autogel, but erroneously received placebo.) | 56 (One subject was randomised to receive lanreotide Autogel, but erroneously received placebo.)
Completed | 45 (Received 4 DB study injections AND continued to IOL phase OR) | 34 (had diary data at least up to day 21 after 4th dose, regardless of missing diary data before day 21.)
Not Completed | 14 | 22
Not completed — Early Roll Over (ERO) to IOL phase | 11 | 12
Not completed — Adverse Event | 1 | 2
Not completed — Subject Decision | 1 | 5
Not completed — Sponsor Decision | 0 | 1
Not completed — Disease Progression | 1 | 1
Not completed — Started Nonprotocol Radiation therapy | 0 | 1
Period: IOL Phase
Arm/Group | Lanreotide Autogel (Somatuline Depot) 120 mg | Placebo
Started | 56 | 46 (Includes 1 subject listed as completing and withdrawing from the DB phase due to brain radiation)
Completed | 43 | 37
Not Completed | 13 | 9
Not completed — Adverse Event | 1 | 1
Not completed — Subject Decision | 4 | 3
Not completed — Physician Decision | 3 | 2
Not completed — Sponsor Decision | 1 | 0
Not completed — Disease Progression | 2 | 1
Not completed — Subject Consumed Prohibited Medication | 1 | 0
Not completed — Peptide Receptor Radionuclide Therapy | 0 | 1
Not completed — Other | 1 | 0
Not completed — Brain radiation | 0 | 1
Period: LTOLE Phase
Arm/Group | Lanreotide Autogel (Somatuline Depot) 120 mg | Placebo
Started | 32 (24 subjects from IOL did not enter LTOLE (11 completed IOL, 13 did not complete IOL).) | 25 (20 subjects from IOL did not enter LTOLE (12 completed IOL, 8 did not complete IOL).)
Completed | 17 | 8
Not Completed | 15 | 17
Not completed — Adverse Event | 7 | 3
Not completed — Subject decision | 0 | 5
Not completed — Physician Decision | 4 | 1
Not completed — Sponsor decision | 2 | 1
Not completed — Disease Progression | 2 | 5
Not completed — Tumour Progression of Hepatic Metastases | 0 | 1
Not completed — Proton Pump Inhibitor Dose Adjusted | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: All randomised subjects (regardless of whether the subjects received or adhered to the allocated treatment group). Subjects from the ITT population were analysed under the randomised treatment group.
Groups:
- Lanreotide Autogel (Somatuline Depot) 120 mg: Deep s.c. injections of lanreotide Autogel 120 mg every 4 weeks (±3 days) for 16 weeks (DB phase). Subjects then received deep s.c. injections of lanreotide Autogel 120 mg every 4 weeks for 32 weeks in the IOL phase and further deep s.c. injections with lanreotide Autogel every 4 weeks in the LTOLE phase. Intent-to-treat (ITT) population: All randomised subjects (regardless of whether the subjects received or adhered to the allocated treatment group). Subjects from the ITT population were analysed under the randomised treatment group.
- Total: Total of all reporting groups
Arm/Group | Lanreotide Autogel (Somatuline Depot) 120 mg | Placebo | Total
Number analyzed (Participants) | 59 | 56 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (10.6) | 59.3 (11.6) | 58.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 35 | 67
  Male | 27 | 21 | 48
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 6 | 3 | 9
  Black/African American | 2 | 3 | 5
  White | 44 | 44 | 88
  Multi race | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days With Subcutaneous Octreotide as Rescue Medication
Description: Use of s.c. octreotide required to control symptoms associated with carcinoid syndrome, measured as the percentage of days that s.c. octreotide was used as rescue medication, based on subject Interactive Voice Response System (IVRS) or Interactive Web Response System (IWRS) diary records.
Time Frame: 16-week DB phase
Population: ITT population: All randomised subjects (regardless of whether the subjects received or adhered to the allocated treatment group). Subjects from the ITT population were analysed under the randomised treatment group.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of days
Groups:
- Lanreotide Autogel (Somatuline Depot) 120 mg: Deep s.c. injections of lanreotide Autogel 120 mg every 4 weeks (±3 days) for 16 weeks (DB phase).
- Placebo: Deep s.c. injections of placebo every 4 weeks (±3 days) for 16 weeks (DB phase).
Arm/Group | Lanreotide Autogel (Somatuline Depot) 120 mg | Placebo
Number analyzed (Participants) | 59 | 56
Percentage of days | 33.72 [25.02 to 42.42] | 48.49 [39.57 to 57.40]
Statistical Analysis 1: Comparison: Lanreotide Autogel (Somatuline Depot) 120 mg vs Placebo; Test type: Superiority or Other; p = 0.0165, ANCOVA; This analysis does not include any imputation for the early roll over subjects

2. Secondary Outcome: Average Frequency of Diarrhoea Events (Per Day) Based on Subject Diary Records.
Time Frame: 16-week DB phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of events per day
Arm/Group | Lanreotide Autogel (Somatuline Depot) 120 mg | Placebo
Number analyzed (Participants) | 59 | 56
Number of events per day | 1.56 (1.83) | 1.35 (1.45)
Statistical Analysis 1: Comparison: Lanreotide Autogel (Somatuline Depot) 120 mg vs Placebo; Test type: Superiority or Other; p = 0.2544, ANCOVA; ANCOVA included treatment group and 2 stratification variables at randomisation as factors and average frequency of diarrhoea per day during Screening

3. Secondary Outcome: Average Frequency of Flushing Events (Per Day) Based on Subject Diary Records.
Time Frame: 16-week DB phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of events per day
Arm/Group | Lanreotide Autogel (Somatuline Depot) 120 mg | Placebo
Number analyzed (Participants) | 59 | 56
Number of events per day | 0.92 (1.45) | 1.75 (2.26)

4. Secondary Outcome: Percentage of Days of Use of Other Rescue Medication
Description: Usage of other concomitant rescue medications for diarrhoea and/or flushing events, measured as the percentage of days that the medications were used as rescue medication based on subject IVRS/IWRS diary records. Subjects were required to record the use and dose of s.c. octreotide, if any, as well as the use of other concomitant rescue medications (e.g. loperamide 2 mg tabs, and/or tincture of opium).
Time Frame: 16-week DB phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Lanreotide Autogel (Somatuline Depot) 120 mg | Placebo
Number analyzed (Participants) | 59 | 56
Percentage of days | 8.86 (19.34) | 6.25 (17.48)

5. Secondary Outcome: Proportion of Subjects Who Rolled Over Into the IOL Phase Before Completing the DB Phase of the Study
Description: Subjects who rolled over early were those who received less than four DB injections before receiving the first IOL injection.
Time Frame: 16-week DB phase
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Lanreotide Autogel (Somatuline Depot) 120 mg | Placebo
Number analyzed (Participants) | 59 | 56
Percentage of subjects | 18.6 | 21.4

6. Secondary Outcome: Changes From Baseline in "Global Health Status/Quality of Life (QoL)" Score (Based on Items 29 and 30 of the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire [EORTC-QLQ] C30)
Description: Baseline is defined as the last non-missing observation obtained prior to the initiation of study treatment.
  Q29 and Q30 range from 1 (Very poor) to 7 (Excellent) with 1 being worst case and 7 the most favourable answer. Scores were derived according to the rules contained within the EORTC scoring manual. All of the scores range in score from 0 to 100. A high score for global health status/QoL represents high QoL. The principle for scoring the scale is: Estimate the average of the items (I1, I2, ..., In) that contribute to the scale; this is the raw score. Raw score = RS = (I1 + I2 +…+ In)/n.
  For global health status/QoL: Score = {(RS - 1)/range} x 100, where range is the difference between the maximum possible value of RS and the minimum possible value of RS.
Time Frame: Baseline and Week 12 of DB phase
Population: ITT population: All randomised subjects (regardless of whether the subjects received or adhered to the allocated treatment group); n=number of subjects taken into account for the analysis. Only the observed data are used in the calculation. The missing data are excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lanreotide Autogel (Somatuline Depot) 120 mg | Placebo
Number analyzed (Participants) | 48 | 34
Units on a scale | 4.17 (14.18) | -1.72 (18.21)

7. Secondary Outcome: Changes From Baseline in "Gastrointestinal (G.I). Symptoms" Subscore (Based on Items Q34, Q35, Q36, Q37 and Q38 of EORTC G.I. Neuroendocrine Tumour [NET] 21]
Description: Baseline is defined as the last non-missing observation obtained prior to the initiation of study treatment.
  The QLQ-G.I.NET21 questionnaire contains 21 single items (Q31 to Q51) which are supplemental items to the EORTC QLQ-C30 questionnaire. Q31 to Q51 range from 1 to 4 with 1 being the most favourable answer and 4 the worst case (1 = Not at all, 2 = A little, 3 = Quite a bit, 4 = Very much). Based on these items the scores were generated. All of the scores range in score from 0 to 100. A high score for a symptom scale represents a high level of symptomatology. The principle for scoring the scale is: Estimate the average of the items (I1, I2, ..., In) that contribute to the scale; this is the raw score. RS = (I1 + I2 +…+ In)/n.
  For symptom scales: Score = {(RS - 1)/range} x 100, where range is the difference between the maximum possible value of RS and the minimum possible value of RS.
Time Frame: Baseline and Week 12 of DB phase
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lanreotide Autogel (Somatuline Depot) 120 mg | Placebo
Number analyzed (Participants) | 48 | 33
Units on a scale | -4.06 (12.80) | 0.10 (13.83)

8. Secondary Outcome: Changes From Baseline in QoL in "Endocrine Symptoms" Subscore (Assessed Based on Items Q31, Q32 and Q33 Using EORTC QLQ-G.I.NET-21 Questionnaires)
Description: as for outcome 7
Time Frame: Baseline and Week 12 of DB phase
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lanreotide Autogel (Somatuline Depot) 120 mg | Placebo
Number analyzed (Participants) | 48 | 33
Units on a scale | -6.83 (18.98) | -2.69 (22.23)

9. Secondary Outcome: Absolute Changes From Baseline in Biochemical Markers (Plasma Chromogranin A [CgA])
Description: Baseline is defined as the last non-missing observation obtained prior to the initiation of study treatment.
Time Frame: Baseline and Week 12 of DB phase
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Lanreotide Autogel (Somatuline Depot) 120 mg | Placebo
Number analyzed (Participants) | 41 | 28
μg/L | 1125.8 (12579.4) | 801.5 (2294.0)

10. Secondary Outcome: Absolute Changes From Baseline in Biochemical Markers (Urinary 5-hydroxyindoleacetic Acid [5-HIAA])
Description: Baseline is defined as the last non-missing observation obtained prior to the initiation of study treatment.
Time Frame: Baseline and Week 12 of DB phase
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: μmol/day
Arm/Group | Lanreotide Autogel (Somatuline Depot) 120 mg | Placebo
Number analyzed (Participants) | 39 | 27
μmol/day | -201.4 (1009.9) | 36.3 (142.3)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time the subject signed informed consent to the exit visit (up to 16 weeks of DB phase, 32 weeks of IOL phase and every 4 subsequent weeks in the LTOLE phase until at least 2 years after the last subject completed the IOL phase or when marketing approval for the treatment of symptoms of carcinoid syndrome was obtained [whichever occurred first]).
Description: Safety population: All randomised subjects who received at least 1 injection of study treatment; subjects were analysed under the actual treatment received. For placebo group (DB phase) n=57 as 1 subject was randomised to lanreotide Autogel but erroneously received placebo.
  Treatment-emergent AEs (TEAEs) reported in the IOL or LTOLE phases are AEs that were either not present or were of moderate or severe intensity prior to the first dose of lanreotide Autogel during that phase.
Groups:
- Lanreotide Autogel (Somatuline Depot) 120 mg (DB Phase): Deep s.c. injections of lanreotide Autogel 120 mg every 4 weeks (±3 days) for 16 weeks (DB phase). Subjects then received deep s.c. injections of lanreotide Autogel 120 mg every 4 weeks for 32 weeks in the IOL phase and further deep s.c. injections with lanreotide Autogel every 4 weeks in the LTOLE phase.
- Placebo (DB Phase): Deep s.c. injections of placebo every 4 weeks (±3 days) for 16 weeks (DB phase). Subjects then received deep s.c. injections of lanreotide Autogel 120 mg every 4 weeks for 32 weeks in the IOL phase and further deep s.c. injections with lanreotide Autogel every 4 weeks in the LTOLE phase.
- Lanreotide Autogel (Somatuline Depot) 120 mg (IOL Phase): All 101 subjects in the IOL phase received deep s.c. injections of lanreotide Autogel 120 mg every 4 weeks for 32 weeks (56 and 45 of these subjects received treatment with lanreotide Autogel and placebo, respectively, during the DB phase).
- Lanreotide Autogel (Somatuline Depot) 120 mg (LTOLE Phase): All 57 subjects in the LTOLE phase received further deep s.c. injections of lanreotide Autogel 120 mg every 4 weeks (32 and 25 of these subjects received treatment with lanreotide Autogel and placebo, respectively, during the DB phase).
Arm/Group | Lanreotide Autogel (Somatuline Depot) 120 mg (DB Phase) | Placebo (DB Phase) | Lanreotide Autogel (Somatuline Depot) 120 mg (IOL Phase) | Lanreotide Autogel (Somatuline Depot) 120 mg (LTOLE Phase)
Serious Adverse Events (participants affected / at risk) | 2/58 | 5/57 | 8/101 | 15/57
Other Adverse Events (participants affected / at risk) | 31/58 | 34/57 | 71/101 | 46/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Autogel (Somatuline Depot) 120 mg (DB Phase) (N=58) | Placebo (DB Phase) (N=57) | Lanreotide Autogel (Somatuline Depot) 120 mg (IOL Phase) (N=101) | Lanreotide Autogel (Somatuline Depot) 120 mg (LTOLE Phase) (N=57)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (3) | 0 (0) | 3 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness permanent (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide Autogel (Somatuline Depot) 120 mg (DB Phase) (N=58) | Placebo (DB Phase) (N=57) | Lanreotide Autogel (Somatuline Depot) 120 mg (IOL Phase) (N=101) | Lanreotide Autogel (Somatuline Depot) 120 mg (LTOLE Phase) (N=57)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (5) | 8 (9) | 4 (5)
Vomiting (Gastrointestinal disorders) | 4 (6) | 2 (2) | 6 (6) | 5 (8)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 7 (7) | 11 (14) | 13 (25)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 7 (9)
Headache (Nervous system disorders) | 7 (7) | 3 (3) | 10 (15) | 5 (7)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 5 (5) | 2 (2)
Fatigue (General disorders) | 2 (2) | 4 (4) | 10 (10) | 9 (14)
Oedema peripheral (General disorders) | 0 (0) | 3 (3) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 5 (6)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 6 (6) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 5 (5) | 8 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 7 (8) | 6 (9)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (7)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 7 (8) | 5 (5)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (4)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (9) | 7 (12)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 9 (9) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 6 (6) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 5 (5) | 4 (5)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 9 (10) | 5 (5)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (5) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (10)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 5 (12)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (2) | 3 (3) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1) | 2 (2) | 6 (9)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4) | 6 (7)

LIMITATIONS AND CAVEATS:
None specified.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
With permission from the Sponsor, each investigator may have published or reported data from their own subjects. The study data in aggregate are the property of the Sponsor and may not be published without permission of the Sponsor. The Sponsor is the final arbitrator of issues relating to the publication or presentation of the aggregate data.